CLINICAL TRIAL: NCT02383992
Title: Comparing the Efficacy of Hydrogen Peroxide Versus Normal Saline in Postoperative Care of Sutured Wounds
Brief Title: Postoperative Care of Sutured Wounds
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Participants never enrolled, study never started.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology-Head and Neck Surgery, and Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU200234
Record Dates: First submitted 2015-03-04; First posted 2015-03-10 (Estimated); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Wound Healing
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydrogen Peroxide (Active Comparator): Post-operative wound will be treated with 3% H2O2 solution, Subjects will also clean the sutured wounds with 3% H2O2 solution or twice daily then dress the wounds with petroleum jelly and a bandage.
  Interventions: Drug: 3% H2O2 solution
- Saline (Active Comparator): Post-operative wound will be treated with 0.9% normal saline. Subjects will also clean the sutured wounds with normal saline twice daily then dress the wounds with petroleum jelly and a bandage.
  Interventions: Drug: 0.9% normal saline

INTERVENTIONS:
Drug: 3% H2O2 solution
  Arms: Hydrogen Peroxide
Drug: 0.9% normal saline
  Arms: Saline

SUMMARY:
The primary objective of this study is to compare the efficacy of hydrogen peroxide versus normal saline in postoperative care of sutured wounds. Subjects will be randomly assigned to standard of care hydrogen peroxide or standard of care normal saline in postoperative care of sutured wounds followed by applying petroleum jelly and sterile gauze bandage. Data will be collected at day 0 and between days 7 to14. Subjects will provide irritation scale rating (0-4) with 0 being none/absent and 4 being severe/extreme.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are undergoing sutured wound after dermatologic procedure.
2. Males and females ages 18-65 years old.
3. Patients who are in good health.
4. Willingness and the ability to understand and provide informed consent and communicate with the investigator/study staff.

Exclusion Criteria:

1. History of keloids or hypertrophic scars.
2. History of bleeding tendency or coagulopathy.
3. Pregnant or lactating or intends to become pregnant in the next 3 months.
4. Active skin disease or skin infection in the treatment area.
5. Unable to understand the protocol or to give informed consent.
6. Any other condition that would, in the professional opinion of the investigator, potentially affect response or participation in the clinical clinical study, or would pose as an unacceptable risk to the subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Irritation scale rating from 1-2 weeks compared to baseline | Baseline and 1-2 weeks
  Subjects will provide irritation scale rating (0-4) with 0 being none/absent and 4 being severe/extreme.

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States